CLINICAL TRIAL: NCT04032886
Title: Does Mechanical Correction Reduce Muscle Stiffness in People With Rounded Shoulder?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, özge ece günaydın, Head of The Physiotherapy and Rehabilitation Department, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/14
Record Dates: First submitted 2019-07-18; First posted 2019-07-25 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Posture
Keywords: kinesio tape; posture; elastography
MeSH Terms: interventions — Athletic Tape; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- classic kinesio tape (Experimental): this group will receive mechanical correction tape with classic tape plus exercise.
  Interventions: Other: kinesio tape; Other: exercise
- performance kinesio tape (Experimental): this group will receive mechanical correction tape with performance tape plus exercise.
  Interventions: Other: kinesio tape; Other: exercise
- control (Other): this group will receive only exercise.
  Interventions: Other: exercise

INTERVENTIONS:
Other: kinesio tape — This is a taping method used for correction of rounded shoulders.
  Other Names: exercise
  Arms: classic kinesio tape; performance kinesio tape
Other: exercise — Exercises include basic postural exercises.

SUMMARY:
The primary aim of this study is to investigate the effect of mechanical correction taping on the stiffness of the upper trapezius and pectoralis minor muscles in patients with rounded shoulder deformity. The secondary aim of our study was to see whether different tape materials affect the application results.

DETAILED DESCRIPTION:
Mechanical correction technique is a highly preferred method among users. Besides its tactical stimulation it serves like a tool helping to reposition the joints.

Here in this study, the investigators aimed to see the secondary effect of the technique on posture. İt is already known that mechanical correction supports the joints and posture but, the question is; by supporting the upright position does it help the extra loaded muscles to release? As the best way to measure the stiffness of the muscles is Elastography, this study will highlight an important issue about correcting posture and regulate muscle loading.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 30 years,
* Sedentary
* Volunteer to enroll in the study,
* To have rounded shoulders,
* To have upper body pain

Exclusion Criteria:

* Professional sports participants
* Musculoskeletal injury during the last 6 months
* Neurologic disorders
* Cervical disc herniation
* To receive physical therapy regarding shoulders in the past 6 months
* Any orthopaedic disorders including impingement, tendinitis, bursitis etc.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postural muscle stiffness is more common in females.
Enrollment: 42 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
change from baseline shearwave elastography stiffness levels to 4 weeks | 4 weeks
  this method will be used to see the stiffness of muscles
change from baseline postural angle degrees to 4 weeks | 4 weeks
  forward head and rounded shoulder positions will be assessed with a smartphone based application.
change from baseline rounded shoulder measurement to 4 weeks | 4 weeks
  this will measure the distance between acromion and the table while the participant is in supine position

SECONDARY OUTCOMES:
change from baseline Penn shoulder scale total score to 4 weeks | 4 weeks
  Originally published in 1999 in Disorders of the Shoulder: Diagnosis and Management, the Penn Shoulder Score assesses patient pain (3 items), satisfaction (1 item), and function (20 items). This is a patient-reported outcome tool and the scores range from 0 to 100 with a score of 100 indicating low pain, high satisfaction, and high function. This is a joint-specific score, which may be useful for individuals with shoulder pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided